CLINICAL TRIAL: NCT05761379
Title: Clinical Study of Low Lever Red Light Therapy With 650nm to Control Myopia Progression in Children
Brief Title: Clinical Study of Light Therapy to Control Myopia Progression in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Airdoc Technology Co., Ltd. (Industry)
Collaborators: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingAirdoc
Record Dates: First submitted 2023-02-03; First posted 2023-03-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Intervention Model Description: Low lever red light therapy with Model : Sky-n1201c at the wavelength of 650nm; 3 minutes illumination for both eyes, administered twice daily at the interview of 4 hours.
  Children in the red light therapy group wore single vision spectacles the entire day and under red light therapy (power, 0.6mW; wavelength, 650nm; Beijing Airdoc MPC Co. Ltd, Beijing, China) twice per day for 3 minutes each session, with at least a 4-hour interval between sessions. There were no specific guidelines for room illumination. After the first measurement session, each child returned for follow-up examinations at 1, 3, and 6 months and completed all the aforementioned examinations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PBM therapy 1 (Experimental): PBM therapy was performed with a low-intensity laser (Airdoc, MPC Co.,Ltd., Beijing, China) with an irradiance of 0.6±0.2 mW, a wavelength of 650 nm±10 nm, and illumination of approximately 400 lux on average. The lighting spot for therapy is a dot. Only one eye will be treated with PBM therapy.
  Interventions: Device: Photobiomodualtion Therapy; Device: Single vision spectacles for correction myopia
- PBM therapy 2 (Experimental): PBM therapy was performed with a low-intensity laser (Airdoc, MPC Co.,Ltd., Beijing, China) with an irradiance of 0.3±0.2 mW, a wavelength of 650 nm±10 nm, and illumination of approximately 400 lux on average. Only one eye will be treated with PBM therapy.
  Interventions: Device: Photobiomodualtion Therapy; Device: Single vision spectacles for correction myopia
- Control (Placebo Comparator): Single vision spectacles correction only.
  Interventions: Device: Single vision spectacles for correction myopia

INTERVENTIONS:
Device: Photobiomodualtion Therapy — low lever light therapy with laser semi-conductor at wavelength of 650nm
  Other Names: Myopia light therapy; Low lever light therapy; Low lever laser therapy; Low intensity red light thearpy
  Arms: PBM therapy 1; PBM therapy 2
Device: Single vision spectacles for correction myopia — Provide the distance best corrected vision acuity of refractive error of myopia for all the groups
  Other Names: Glasseses

SUMMARY:
Low-lever red light therapy (LLLT) has been used to control myopia progression in China for a few years besides amblyopia therapy for a few decades. This study is to test the efficacy of PBM therapy to myopia children as well as to compare two types of PBM therapy to control myopia progression within one month.

DETAILED DESCRIPTION:
LLLT utilized the 650-nm red light to provide sufficient energy to stimulate the tissue without causing damage to the surrounding tissues. And several researchers reported the long-term efficacy of LLLT in slowing the progression of myopia to date. These studies were reported various illumination and irradiance. This study is to test the efficacy of LLLT comparing to the control group as well as to test whether two types of lighting design will be different to the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Grade 1 to grade 9 and age 6 to 16 years (including 6 and 16 years), Sex is not limited;
2. Equivalent sphere (SER): -0.50D ~ -6.00D (including-0.50 and-6.00D);
3. Best corrected vision in one eye under glasses correction: 0.1 log MAR;
4. No strabismus: no more than 15 prism constant dominance strabismus after far and near cover tests;
5. No myopia control measures within the previous 4 weeks: such as orthokeratology lens, gradient lens, double light lens, eye drops for myopia control (such as atropine), myopia defocus glasses, red light for myopia control, other specially designed myopia light treatment instruments or contact lenses for special design to control myopia (such as Misight);

Exclusion Criteria:

1. Any ocular(including constant dominant strabismus with more than 15 prisms) and systemic diseases or abnormalities can significantly affect visual function or promote the progression of myopia;
2. Other interventions for myopia control before 4 weeks before enrollment, For example, orthoplastic lens, gradient lens, dual-light lens, eye drops for myopia control (atropine), myopia defocus glasses, red light therapy devices for myopia control, other specially designed comprehensive treatment devices, myopia, amblyopia, or specially designed contact lenses (such as Misight), etc.
3. Subject participated in other clinical trials within 4 weeks before the enrollment;
4. The investigator for safety reasons or the interests of the patient, Other circumstances in which the patient should not participate in this trial, If suffering from serious heart, liver and kidney disease. -

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in axial length (mm） | at 1-month Follow-up
  Changes of axial length at 1-Month follow-up from baseline with IOLmaster 500
  Axial length measurement at baseline and at follow-up with IOLmaster(Carl Zeiss). Five measurements were taken and averaged. The changes will be calculated by the formula as below: Change in axial length ( mm ) = Axial length value at follow-up baseline

SECONDARY OUTCOMES:
Changes in cycloplegic autorefraction (diopters, D) | at 1-month Follow-up and at baseline
  Objective refraction measured by using Autorefractor. Five measurements are obtained for each eye and the average of spherical equivalence was used for statistical analysis. The measurements will be both with cycloplegia at baseline and at follow-up. The changes in cycloplegic autorefraction are calculated in the mean value of each group.
Changes of choroidal thickness under macular foveal (um) | at 1-month Follow-up and at baseline
  Swept-source optical coherence tomography (OCT) and OCT angiography were used To measure choroidal fovea thickness at baseline and at follow-up. To avoid the effects of circadian rhythm on the results, OCT scanning was performed twice by the same investigator between 8:00 A.M. and 2:00 P.M. at baseline and 1-month follow-up. Two independent skilled professionals measured the sub-foveal choroidal thickness （SFChT) using a linear measurement program during the OCT scan. To increase the visibility of the choroid, the enhanced depth imaging mode was used. We defined the thinnest part of the macula in the image as the fovea. The SFChT was measured from the outermost part of the retinal pigment epithelium to the inner layer of the the choroidoscleral interface.
Changes of cornea power | at 1-month Follow-up and at baseline
  Changes in the central anterior cornea power by the value measured from auto-refraction. The mean values will be recorded as well as the mean values at follow-up of 1 month
Change in retina fovea perfusion density (RFPD, %) | at 1-month Follow-up and at baseline
  Swept-source optical coherence tomography (OCT) angiography is used to measure retina fovea perfusion density (RFPD). The TowardPi OCTA allow for the in vivo visualization of three-dimensional (3-D) vascular networks in the retina and choroid. The OCTA images were acquired by the TowardPi-3D spatial identification algorithm. The retina vessels and choriocapillaris were identified by higher order moments decorrelation algorithm. The medium- and large-sized choroid vessels from Sattler's layer and Haller's layer were visualized by 3D threshold segmentation algorithm. In this study, the retinal and choroidal images were obtained with an area of 18*18 mm centered on the fovea. In addition, for a comprehensive analysis of the macular zone, we adopted the Early Treatment Diabetic Retinopathy Study (ETDRS) grid using the instrument's software which was adjusted for each individual participant's ocular magnification.

CONTACTS AND LOCATIONS:
Overall Officials: Xingtao Zhou, M.D. PhD., Study Chair — Eye & ENT Hospital of Fudan University; Weicun Chen, MD, PhD, Study Director — Eye & ENT Hospital of Fudan University; Meiyan Li, MD, PhD, Study Director — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang W, Lin F, Li M, Wei R, Zhou J, Zhou X. Immediate Effect in the Retina and Choroid after 650 nm Low-Level Red Light Therapy in Children. Ophthalmic Res. 2023;66(1):312-318. doi: 10.1159/000527787. Epub 2022 Oct 31. PMID 36315988
- [Background] Liu G, Li B, Rong H, Du B, Wang B, Hu J, Zhang B, Wei R. Axial Length Shortening and Choroid Thickening in Myopic Adults Treated with Repeated Low-Level Red Light. J Clin Med. 2022 Dec 17;11(24):7498. doi: 10.3390/jcm11247498. PMID 36556114